CLINICAL TRIAL: NCT06459167
Title: Position Intervention to Reduce Hypoxemia in Sedation Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Zhejiang Provincial Tongde Hospital (Other); Shenzhen Second People's Hospital (Other); Zhejiang Provincial People's Hospital (Other); The Sixth Affiliated Hospital of Wenzhou Medical University (Other); Lishui Municipal Central Hospital (Other Government); Ningbo No. 1 Hospital (Other); Zunyi Medical College (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, xiangming fang, Director, Head of Anesthesiology and Critical Care, Principal Investigator, Professor, First Affiliated Hospital of Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Hypoxemia
Record Dates: First submitted 2024-05-24; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Hypoxemia; Sedation Complication; Emergencies; Airway Remodeling
Keywords: position; hypoxemia; sedation; emergency; upper airway
MeSH Terms: conditions — Hypoxia; Emergencies; Airway Remodeling | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): Patients needing sedation for procedure or surgery are assisted into supine position before they were sedated and kept during the procedure.
  Interventions: Other: The position adopted when patients undergoing procedure or surgery
- Group L (Experimental): Patients needing sedation for procedure or surgery are assisted into lateral position before they were sedated and kept the procedure.
  Interventions: Other: The position adopted when patients undergoing procedure or surgery

INTERVENTIONS:
Other: The position adopted when patients undergoing procedure or surgery — For patients requiring sedation for procedures or surgery, they are randomly assigned either to supine position or lateral position before they are sedated, and kept during procedure or surgery.

SUMMARY:
Hypoxemia was defined as an SpO2 of < 90% for any duration. Failure to treat promptly can lead to hypoxemia, which may increase the risks of arrhythmia, nausea and vomiting, and cognitive dysfunction. Studies have shown that body position has a direct impact on respiratory function. In special environments, including outside the operating room where emergency airway management for critically ill and injured patients is needed, or in areas with limited medical resources like remote areas, adopting simple interventions by changing position to maintain patients' respiratory function can be more economical, convenient and safe.

DETAILED DESCRIPTION:
Hypoxemia was defined as an SpO2 of < 90% for any duration. Failure to treat promptly can lead to hypoxemia, which may increase the risks of arrhythmia, nausea and vomiting, and cognitive dysfunction. Studies have shown that body position has a direct impact on respiratory function. In special environments, including outside the operating room where emergency airway management for critically ill and injured patients is needed, or in areas with limited medical resources like remote areas, adopting simple positional interventions to maintain patients' respiratory function can be more economical, convenient and safe. This study aims to conduct a prospective, multicenter, randomized controlled trial to observe the level of patients' oxygen saturation and the occurrence of hypoxemia under different body positions (supine and lateral positions), and its impact on prognosis, providing reliable evidence-based medical evidence for the prevention and treatment of complications in patients requiring airway management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with 18 years or older
2. Without obvious cardiovascular or pulmonary dysfunction
3. Scheduled to undergo procedure or surgery with sedation
4. Signed the informed consent form

Exclusion Criteria:

1. Preexisting bradycardia (heart rate <50 beats/min), hypotension (systolic blood pressure < 80mmHg), or hypoxemia (SpO2 < 90%);
2. Requiring supplemental chronic or intermittent oxygen therapy because of preexisting diseases
3. Preexisting diseases which unable to tolerate reduced SpO2 or Partial pressure of carbon dioxide in artery (PaCO2) diseases, such as severe cardiovascular and cerebrovascular diseases, intracranial hypertension or severe lung diseases;
4. Coagulation disorders or a tendency of nose bleeding;
5. Patients whose body position cannot be altered;
6. Participated in other intervention clinical studies in the past 3 months;
7. Other conditions deemed unsuitable for inclusion by the researcher;
8. Patients and guardians refused to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1752 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The lowest SpO2 | During procedure
  The lowest SpO2 during sedation and procedures
Use of airway interventions | During procedure
  Use of airway interventions including increased inhaled O2, ventilated mask and endotracheal intubation

SECONDARY OUTCOMES:
The onset of when SpO2 dropped below 80% | During procedure
  The onset of when SpO2 reached below 80%
The onset of when SpO2 dropped below 70% | During procedure
  The onset of when SpO2 reached below 70%
The onset of respiratory adverse events | During procedure
  The onset of respiratory adverse events including apnea, laryngospasm, aspiration due to regurgitation
The onset of circulatory adverse events | During procedure
  The onset of circulatory adverse events including hypotension, hypertension, bradycardia, tachycardia, new-onset arrhythmia with hemodynamically stable/instability, cardiac arrest, shock
The onset of gastrointestinal adverse events | During procedure
  The onset of gastrointestinal adverse events including nausea and vomiting, regurgitation
The degree of operator satisfaction | During procedure
  The degree of operator satisfaction regarding the performance, effectiveness, and experience of a procedure. A 10-point scale is used, 0 indicates complete dissatisfaction and 10 indicates complete satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangming Fang, M.D., Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klare P, Huth R, Haller B, Huth M, Weber A, Schlag C, Reindl W, Schmid RM, von Delius S. Patient position and hypoxemia during propofol sedation for colonoscopy: a randomized trial. Endoscopy. 2015 Dec;47(12):1159-66. doi: 10.1055/s-0034-1392329. Epub 2015 Jun 30. PMID 26126161
- [Result] Ababneh O, Bsisu I, El-Share' AI, Alrabayah M, Qudaisat I, Alghanem S, Khreesha L, Ali AM, Rashdan M. Awake Nasal Fiberoptic Intubation in Lateral Position for Severely Obese Patients with Anticipated Difficult Airway: A Randomized Controlled Trial. Healthcare (Basel). 2023 Oct 24;11(21):2818. doi: 10.3390/healthcare11212818. PMID 37957962
- [Result] Edmark L, Kostova-Aherdan K, Enlund M, Hedenstierna G. Optimal oxygen concentration during induction of general anesthesia. Anesthesiology. 2003 Jan;98(1):28-33. doi: 10.1097/00000542-200301000-00008. PMID 12502975
- [Result] Semler MW, Janz DR, Russell DW, Casey JD, Lentz RJ, Zouk AN, deBoisblanc BP, Santanilla JI, Khan YA, Joffe AM, Stigler WS, Rice TW; Check-UP Investigators( *); Pragmatic Critical Care Research Group. A Multicenter, Randomized Trial of Ramped Position vs Sniffing Position During Endotracheal Intubation of Critically Ill Adults. Chest. 2017 Oct;152(4):712-722. doi: 10.1016/j.chest.2017.03.061. Epub 2017 May 6. PMID 28487139
- [Result] Wahdan AS, El-Refai NAR, Omar SH, Abdel Moneem SA, Mohamed MM, Hussien MM. Endotracheal intubation in patients undergoing open abdominal surgery in the lateral position: a comparison between the intubating video stylet and fiberoptic intubating bronchoscopy. Korean J Anesthesiol. 2021 Jun;74(3):234-241. doi: 10.4097/kja.20384. Epub 2020 Oct 19. PMID 33070582
- [Result] Leeb G, Auchus I, Law T, Bickler P, Feiner J, Hashi S, Monk E, Igaga E, Bernstein M, Chou YC, Hughes C, Schornack D, Lester J, Moore K Jr, Okunlola O, Fernandez J, Shmuylovich L, Lipnick M. The performance of 11 fingertip pulse oximeters during hypoxemia in healthy human participants with varied, quantified skin pigment. EBioMedicine. 2024 Apr;102:105051. doi: 10.1016/j.ebiom.2024.105051. Epub 2024 Mar 8. PMID 38458110
- [Derived] Ye H, Chu LH, Xie GH, Hua YJ, Lou Y, Wang QH, Xu ZX, Tang MY, Wang BD, Hu HY, Ying J, Yu T, Wang HY, Wang Y, Ye ZJ, Bao XF, Wang MC, Chen LY, Wang XX, Zhang XB, Huang CS, Wang J, Lu YP, Luo FQ, Zhou W, Wang CG, Cheng H, Liu WJ, Luo J, Wu YQ, Li RR, Wang D, Hou LQ, Shi L, Zhang J, Wang K, Pi X, Zhou R, Yang QQ, Wan PL, Li H, Wu SJ, Song SW, Cui P, Shu L, Islam N, Fang XM. Effect of lateral versus supine positioning on hypoxaemia in sedated adults: multicentre randomised controlled trial. BMJ. 2025 Aug 19;390:e084539. doi: 10.1136/bmj-2025-084539. PMID 40829895